CLINICAL TRIAL: NCT01219049
Title: L-Tyrosine Supplementation in Patients With Fibromyalgia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to FDA comments, changes required unavailable resources. There are no results for this study.
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09-1144
Record Dates: First submitted 2010-10-08; First posted 2010-10-13 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Fibromyalgia
Keywords: Diet; Fibromyalgia; Pain; Drug; Amino-acid; Fatigue
MeSH Terms: conditions — Fibromyalgia; Pain; Fatigue | interventions — Tyrosine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tyrosine 1000 mg / day (Experimental): Patients receive 1000 mg tyrosine per day.
  Interventions: Drug: Tyrosine
- Tyrosine 2000 mg / day (Experimental): Patients receive 2000 mg tyrosine per day.
  Interventions: Drug: Tyrosine
- Placebo (Placebo Comparator): Patients receive placebo daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tyrosine — 1000 mg / day
  Arms: Tyrosine 1000 mg / day
Drug: Tyrosine — 2000 mg / day
  Arms: Tyrosine 2000 mg / day
Drug: Placebo — Placebo daily
  Arms: Placebo

SUMMARY:
Patients in the study, who have a diagnosis of fibromyalgia, will be randomly assigned to take the amino acid L-tyrosine or placebo (blank pill) for 3 weeks. They will fill out questionnaires about their symptoms and see if they have any improvement. The investigators hypothesis is that taking tyrosine will help alleviate the symptoms of fibromyalgia.

DETAILED DESCRIPTION:
Fibromyalgia is a chronic pain syndrome with few treatment options available. The amino-acid L-tyrosine is the precursor for norepinephrine in the central nervous system (CNS). Norepinephrine in the CNS has important roles in pain and mood modulation and descending inhibition of pain pathways. By giving the precursor L-tyrosine in high doses we believe that we can increase levels of norepinephrine in the CNS. To study this question we designed a randomized blinded pilot study of 30 patients. Patients are randomly assigned to one of 3 groups (placebo, tyrosine 1000mg/day, and tyrosine 2000mg/day.) for 3 weeks. Patients then complete the Brief Pain Inventory (BPI) daily and the Fibromyalgia impact questionnaire (FIQ) on day 1 and day 21. Patients also complete a drug diary. They are monitored weekly for progress during the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of fibromyalgia
* Pain greater than 4/10
* Age greater than 18

Exclusion Criteria:

* Pregnant
* Age less than 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Pain Score | daily for 21 days
FIQ Score | Day 1
FIQ Score | Day 21

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Mazzeffi, MD, MPH, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States